CLINICAL TRIAL: NCT03947710
Title: Acute Effect of Protein Intake During Dialysis on Intradialytic Blood Pressure, 24-hour Ambulatory Blood Pressure and Arterial Stiffness Indices in Maintenance Hemodialysis Patients.
Brief Title: Effect of Protein Intake During Hemodialysis on Blood Pressure and Arterial Stiffness Indices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Vaios Vasileios, Vaios Vasileios, Resident in Nephrology, Department of Nephrology and Hypertension, AHEPA University Hospital, Aristotle University Of Thessaloniki, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MedAuth2
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: End Stage Renal Disease; Hypotension During Dialysis; Protein Malnutrition; Arterial Sclerosis
MeSH Terms: conditions — Kidney Failure, Chronic; Kwashiorkor; Arteriosclerosis

STUDY DESIGN:
Intervention Model Description: Open label, randomized, cross-over clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-protein meals (Experimental): Patients with End Stage Renal disease on maintenance hemodialysis will consume high protein meals during their dialysis sessions for one week.
  Interventions: Other: High-protein meals
- Low-protein meals (Experimental): Patients with End Stage Renal disease on maintenance hemodialysis will consume low protein meals during their dialysis sessions for one week
  Interventions: Other: Low- protein meals
- No meals (Experimental): Patients with End Stage Renal disease on maintenance hemodialysis will not consume meals during their dialysis sessions for one week
  Interventions: Other: No meals

INTERVENTIONS:
Other: High-protein meals — Patients on maintenance hemodialysis will consume high protein meals during dialysis for one week (3 dialysis sessions)
  Arms: High-protein meals
Other: Low- protein meals — Patients on maintenance hemodialysis will consume low protein meals during dialysis for one week (3 dialysis sessions)
  Arms: Low-protein meals
Other: No meals — Patients on maintenance hemodialysis will not consume meals during dialysis for one week (3 dialysis sessions)
  Arms: No meals

SUMMARY:
Open label, randomized, cross-over clinical study comparing the acute effect of high versus low protein meals during dialysis on intradialytic blood pressure, 24-hour ambulatory blood pressure and arterial stiffness indices on maintenance hemodialysis patients.

DETAILED DESCRIPTION:
A series of demographic, anthropometric and clinical data will be collected prior to enrollment. The intervention will last 3 consecutive weeks. Eligible subjects will be randomised to one group (high or low protein meals during dialysis) for one week (3 dialysis sessions). Second week will be a wash out period (patients will not consume meals during dialysis) and during the third week randomised subjects will cross over to the other study group. Every meal will provide 1/3 of daily recommended energy and protein intake (35 kcal/kg body weight/day, 0.7 gr protein/kg body weight/day for low protein meals and 1.5 gr protein/kg body weight/day for high protein meals). All the meals will be prepared in the hospital's kitchen and will be personalized to each patient's preferences. The meal will be given one hour after the start of the session and should be consumed completely during dialysis.

Patients will be evaluated for the following parameters during their midweek dialysis session:

1. Intradialytic blood pressure
2. 24-hour ambulatory blood pressure
3. Arterial stiffness indices (Central Aortic blood pressure, Pulse Wave Velocity, Augmentation Index)
4. Hemodialysis adequacy
5. Nutritional status

Intradialytic blood pressure, 24-hour ambulatory blood pressure and arterial stiffness indices will be evaluated with the use of the brachial cuff-based oscillometric device Mobil-O-Graph NG (IEM, Stolberg, Germany). Urea reduction ratio (URR) and Kt/V (standard and equilibrated) will be used as measures for dialysis adequacy. Possible changes in patients nutritional status will be assessed using the Malnutrition-Inflammation Score (MIS).

ELIGIBILITY:
Inclusion Criteria:

* Patients to have provided informed written consent
* Patients undergoing maintenance hemodialysis for at least 3 months prior to enrollment
* Ability to self-ingest food during the dialysis session

Exclusion Criteria:

* History of malignancy or any other clinical condition associated with very poor prognosis
* Hospitalization for acute myocardial infarction, unstable angina or acute ischemic stroke within the 3 previous months
* Patients receiving parenteral nutrition
* Body mass index (BMI) of >40 kg/m2
* Bilateral functioning or non-functioning arteriovenous fistula (AVF) and/or arteriovenous graft (AVG) used as dialysis access
* Patients with major amputations (eg lower limbs)
* Women during pregnancy or lactation
* Patients with unsuccessful 24-hour ambulatory recording of blood pressure with Mobil-O-Graph device, in accordance with the current European Society of Hypertension Guidelines.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Effect of meal versus no meal consumption during hemodialysis on intradialytic blood pressure | 3 weeks
  Meal consumption is expected to lower intradialytic blood pressure and increase hypotensive events during hemodialysis. Intradialytic blood pressure will be evaluated with the use of the brachial cuff-based oscillometric device Mobil-O-Graph NG (IEM, Stolberg, Germany) during the midweek dialysis session.
Effect of high versus low protein meal consumption during dialysis on intradialytic blood pressure | 3 weeks
  High protein meals are expected to affect less intradialytic blood pressure than low protein meals. Intradialytic blood pressure will be evaluated with the use of the brachial cuff-based oscillometric device Mobil-O-Graph NG (IEM, Stolberg, Germany) during the midweek dialysis session.

SECONDARY OUTCOMES:
Effect of high versus low protein meal consumption during dialysis on 24-hour ambulatory blood pressure | 3 weeks
  24-hour blood pressure will be evaluated with the use of the brachial cuff-based oscillometric device Mobil-O-Graph NG (IEM, Stolberg, Germany). Measurement of 24-hour ambulatory blood pressure will start at the beginning of the midweek dialysis session for each group (high versus low protein meals during dialysis).
Effect of high versus low protein meal consumption during dialysis on Pulse Wave Velocity | 3 weeks
  Pulse Wave Velocity will be measured for each group (high versus low protein meals) during the midweek dialysis session using the brachial cuff-based oscillometric device Mobil-O-Graph NG (IEM, Stolberg, Germany).
Effect of high versus low protein meal consumption during dialysis on Augmentation Index | 3 weeks
  Augmentation Index will be measured for each group (high versus low protein meals) during the midweek dialysis session using the brachial cuff-based oscillometric device Mobil-O-Graph NG (IEM, Stolberg, Germany).
Effect of high versus low protein meals during dialysis on hemodialysis adequacy. | 3 weeks
  Hemodialysis adequacy will be calculated for each patient group (high versus low protein meals) using the Urea reduction ratio (URR) and Kt/V (standard and equilibrated) for the midweek dialysis session.
Effect of high versus low protein meals during dialysis on patients nutritional status | 3 weeks
  Nutritional status will be calculated for each group (high versus low protein meals) using the Malnutrition-Inflammation Score (MIS). The Malnutrition-Inflamation score (MIS) is composed of 10 components which include: dry weight change over the last 3-6 months, current dietary intake, gastrointestinal symptoms, functional capacity (nutritionally related functional impairment), co-morbidity (including number of years on dialysis), decreased fat stores or loss of subcutaneous fat on physical examination (below eyes, triceps, biceps, chest), signs of muscle wasting (temple, clavicle, scapula, ribs, quadriceps, knee, interosseous), body mass index calculation, serum albumin levels, and serum total iron binding capacity. Each component of the MIS has 4 levels of severity, from 0 (normal) to 3 (severely abnormal). The sum of all 10 MIS components can range from 0 (normal) to 30 (severely malnourished); higher score reflects a more severe degree of malnutrition and inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Vassilios Liakopoulos, MD, PhD, Study Chair — Department of Medicine, Aristotle University of Thessaloniki; Elena Fotiadou, Study Director — Department of Nutrition and Dietetics, AHEPA University Hospital, Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Select A State/Province, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caglar K, Fedje L, Dimmitt R, Hakim RM, Shyr Y, Ikizler TA. Therapeutic effects of oral nutritional supplementation during hemodialysis. Kidney Int. 2002 Sep;62(3):1054-9. doi: 10.1046/j.1523-1755.2002.00530.x. PMID 12164890
- [Background] Burrowes JD, Larive B, Cockram DB, Dwyer J, Kusek JW, McLeroy S, Poole D, Rocco MV; Hemodialysis (HEMO) Study Group. Effects of dietary intake, appetite, and eating habits on dialysis and non-dialysis treatment days in hemodialysis patients: cross-sectional results from the HEMO study. J Ren Nutr. 2003 Jul;13(3):191-8. doi: 10.1016/s1051-2276(03)00069-4. PMID 12874743
- [Background] Rhee CM, You AS, Koontz Parsons T, Tortorici AR, Bross R, St-Jules DE, Jing J, Lee ML, Benner D, Kovesdy CP, Mehrotra R, Kopple JD, Kalantar-Zadeh K. Effect of high-protein meals during hemodialysis combined with lanthanum carbonate in hypoalbuminemic dialysis patients: findings from the FrEDI randomized controlled trial. Nephrol Dial Transplant. 2017 Jul 1;32(7):1233-1243. doi: 10.1093/ndt/gfw323. PMID 27659126
- [Background] Jansen RW, Lipsitz LA. Postprandial hypotension: epidemiology, pathophysiology, and clinical management. Ann Intern Med. 1995 Feb 15;122(4):286-95. doi: 10.7326/0003-4819-122-4-199502150-00009. PMID 7825766
- [Background] Choi MS, Kistler B, Wiese GN, Stremke ER, Wright AJ, Moorthi RN, Moe SM, Hill Gallant KM. Pilot Study of the Effects of High-Protein Meals During Hemodialysis on Intradialytic Hypotension in Patients Undergoing Maintenance Hemodialysis. J Ren Nutr. 2019 Mar;29(2):102-111. doi: 10.1053/j.jrn.2018.06.002. Epub 2018 Aug 11. PMID 30107974
- [Background] Kistler B, Benner D, Burgess M, Stasios M, Kalantar-Zadeh K, Wilund KR. To eat or not to eat-international experiences with eating during hemodialysis treatment. J Ren Nutr. 2014 Nov;24(6):349-52. doi: 10.1053/j.jrn.2014.08.003. Epub 2014 Oct 22. PMID 25443543
- [Background] Sarafidis PA, Georgianos PI, Karpetas A, Bikos A, Korelidou L, Tersi M, Divanis D, Tzanis G, Mavromatidis K, Liakopoulos V, Zebekakis PE, Lasaridis A, Protogerou AD. Evaluation of a novel brachial cuff-based oscillometric method for estimating central systolic pressure in hemodialysis patients. Am J Nephrol. 2014;40(3):242-50. doi: 10.1159/000367791. Epub 2014 Oct 11. PMID 25322847
- [Background] San Juan Miguelsanz M, Pilar SM, Santos de Pablos MR. Reduction of Kt/V by food intake during haemodialysis. EDTNA ERCA J. 2001 Jul-Sep;27(3):150-2. doi: 10.1111/j.1755-6686.2001.tb00165.x. PMID 11868999
- [Background] Borzou SR, Mahdipour F, Oshvandi K, Salavati M, Alimohammadi N. Effect of Mealtime During Hemodialysis on Patients' Complications. J Caring Sci. 2016 Dec 1;5(4):277-286. doi: 10.15171/jcs.2016.029. eCollection 2016 Dec. PMID 28032072
- [Background] Bossola M, Luciani G, Rosa F, Tazza L. Appetite and gastrointestinal symptoms in chronic hemodialysis patients. J Ren Nutr. 2011 Nov;21(6):448-54. doi: 10.1053/j.jrn.2010.09.003. Epub 2011 Jan 15. PMID 21239186
- [Background] Sherman RA, Torres F, Cody RP. Postprandial blood pressure changes during hemodialysis. Am J Kidney Dis. 1988 Jul;12(1):37-9. doi: 10.1016/s0272-6386(88)80069-6. PMID 3389352
- [Background] Heymsfield SB, McManus C, Smith J, Stevens V, Nixon DW. Anthropometric measurement of muscle mass: revised equations for calculating bone-free arm muscle area. Am J Clin Nutr. 1982 Oct;36(4):680-90. doi: 10.1093/ajcn/36.4.680. PMID 7124671
- [Background] Frisancho AR. New norms of upper limb fat and muscle areas for assessment of nutritional status. Am J Clin Nutr. 1981 Nov;34(11):2540-5. doi: 10.1093/ajcn/34.11.2540. PMID 6975564
- [Background] Durnin JV, Womersley J. Body fat assessed from total body density and its estimation from skinfold thickness: measurements on 481 men and women aged from 16 to 72 years. Br J Nutr. 1974 Jul;32(1):77-97. doi: 10.1079/bjn19740060. No abstract available. PMID 4843734
- [Background] Malindretos P, Sarafidis P, Spaia S, Sioulis A, Zeggos N, Raptis V, Kitos V, Koronis C, Kabouris C, Zili S, Grekas D. Adaptation and validation of the Kidney Disease Quality of Life-Short Form questionnaire in the Greek language. Am J Nephrol. 2010;31(1):9-14. doi: 10.1159/000252926. Epub 2009 Oct 26. PMID 19864884
- [Background] Agarwal R, Georgianos P. Feeding during dialysis-risks and uncertainties. Nephrol Dial Transplant. 2018 Jun 1;33(6):917-922. doi: 10.1093/ndt/gfx195. PMID 28633456